CLINICAL TRIAL: NCT02683460
Title: Comparison of Clinical Results of Patella Resurfacing Versus Patellar Retention Under Subvastus Approach in Total Knee Arthroplasty: A Randomized, Controlled, Double-Blind Trial
Brief Title: Patellar Resurfacing Under Subvastus Approach in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Patella resurfacing
Record Dates: First submitted 2016-02-04; First posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Osteoarthritis, Patella Resurfacing
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- patella resurfacing group (Experimental): Procedure: Patellar component Resurfacing with onlay technique
  Interventions: Procedure: Patella resurfacing
- patella retention (Active Comparator): Procedure: patellar retention Trimming of osteophytes when appropriate
  Interventions: Procedure: Patella retention

INTERVENTIONS:
Procedure: Patella resurfacing
  Arms: patella resurfacing group
Procedure: Patella retention
  Arms: patella retention

SUMMARY:
This study aims to compare the clinical results of patella resurfacing or not under subvastus approach in total knee arthroplasty. Even though the excellent results of total knee arthroplasty(TKA), there is persistent controversy over whether or not to replace the patella. Anterior knee pain continued to be a unsolved problem of TKA patients. Some surgeons always performed patella resurfacing during total knee arthroplasty but the others didn't do that. It's up to surgeon's preference. There were several studies of patellar resurfacing or not in TKA. But previous studies almost have been done under other approach, not a subvastus approach.

This study prospectively randomized patients receiving bilateral TKA with patellar resurfacing or not in each knee. Patients preference and clinical results was investigated in both knee of same patients who received patellar resurfacing or not during minimum 2 year follow up.

DETAILED DESCRIPTION:
The primary objective of this work was to compare pain, stiffness and function between groups at minimum 2 year postoperatively. Secondarily, we compared pain, patient preference at minimum 2 year postoperatively. The investigators hypothesized that there would be no difference between the two groups of subjects in the measured outcomes.

Patients receiving TKA were prospectively enrolled before surgery and randomized intraoperatively to either receive patella replacement or not in both knee of same patients. Subjects were assessed pre-operatively and at 6 months, 1, 2 years postoperatively for pain, function, and stiffness using a disease-specific (Western Ontario and McMaster Osteoarthritis Index [WOMAC]) . Other measurements like Knee Society score, Feller's score, Patient satisfaction (VAS) also checked pre-operatively and at 6 months, 1, 2 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients for total knee arthroplasty
* Having medicare insurance

Exclusion Criteria:

* Patients who are not able to cooperate
* Serious deformity (not suitable for a standard TKA prosthesis)
* Patellar thickness less than 18 mm
* Prior operation involving the extensor mechanism
* Rheumatoid arthritis
* Severe medical disability limiting the ability to walk
* Revision surgery
* Knees with predominantly patellofemoral arthrosis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
WOMAC (Western Ontario and McMaster University Arthritis Index) pain scale | Change from preoperative score to postoperative 2 years
Knee Society score | Change from preoperative score to postoperative 2 years

SECONDARY OUTCOMES:
Feller's score | Change from preoperative score to postoperative 2 years
Patients satisfaction using Visual Analog Score for pain | Change from preoperative score to postoperative 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yong In, MD, PhD, Study Chair — the Catholic Univerisity of Korea Seoul St Mary's hospital